CLINICAL TRIAL: NCT03627325
Title: Differences in Surgical Risk Evaluation by Surgical Risk Calculator, Residents and Senior Anesthesiologists
Brief Title: The Difference in Preoperative Evaluation That is Given by a Senior Physician, a Specialist, and a Computer Program
Acronym: ACS
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Ronen Ohad, Director Head and Neck Surgery Unit, Western Galilee Hospital-Nahariya
Other Study IDs: NHR-14-OR-0094
Record Dates: First submitted 2018-07-25; First posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients who are scheduled for any surgical procedure — looking for correlation for estimating the complications between the anesthesiologists and the computerized method.

SUMMARY:
There is an increasing need and interest in being able to empirically estimate customized, patient-specific risks for virtually all surgical operations in a user-friendly format.

The ACS (American College of Surgeons) surgical risk calculator is a decision-support tool based on reliable multi institutional clinical data, which can be used to estimate the risks of most operations.1 The aim of this study is to compare the assessment provided by the The ACS Surgical Risk Calculator with the assessment provided by a senior and a resident anesthesiologist, and by that comparison to establish the need for the ACS calculator

DETAILED DESCRIPTION:
Understanding the risks of surgery is clearly important for both patients and surgeons in the shared decision making process. Informed consent requires that patients have a thorough understanding of the potential risks of surgery. Moreover, clinicians and patients also need information regarding surgical risks in order to make decisions on the type of operation or whether surgery should be performed at all.

Therefore, there is a need to discuss the risks derived empirically with a specific patient before any action to guide both surgical decision-making and informed consent.

However, predicting postoperative risks and identifying patients at a higher risk of adverse events have traditionally been based on individual surgeon experience and augmented by published rates in the literature, either from single institution studies or clinical trials. Unfortunately, these estimates are typically not specific to an individual Patient's risk factors. The ACS (American College of Surgeons) Surgical Risk Calculator estimates the chance of an unfavorable outcome (such as a complication or death) after surgery. The risk is estimated based upon information the patient gives to the healthcare provider about prior health history. The estimates are calculated using data from a large number of patients who had a surgical procedure similar to the one the patient may have.

ELIGIBILITY:
Inclusion Criteria:

* Patients candidates for surgery
* Signed informed consent by patient

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for any surgical procedure will be recruited for the study
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2016-08-15 (Actual)

PRIMARY OUTCOMES:
Morbidity for each patient | Each patient is assessed within a week by both physicians and the ACS web-based computer. The trial is scheduled for a whole year.
  Anesthesiologists give their estimation of overall mortality that is compared to that given by the ACS web-based calculator
Morbidity for each patient | Each patient is assessed within a week by both physicians and the ACS web-based computer. The trial is scheduled for a whole year.
  Anesthesiologists give their estimation of different morbidities and that is compared to that given by the ACS web-based calculator

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data available to other researchers